CLINICAL TRIAL: NCT04758429
Title: Validating the Ability for Early Recognition of Worsening Heart Failure by a System Technology of Automated Prediction From Multi-sensor Data: A Prospective, Open-label, Single-arm, International, Multi-center Clinical Study
Brief Title: International Multi-center Study to Validate an Early Warning Algorithm for Worsening Heart Failure
Acronym: VESTA
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chronolife (Industry)
Responsible Party: Sponsor
Other Study IDs: PREDIGMA001
Record Dates: First submitted 2021-02-08; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2021-02

CONDITIONS: Chronic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development or Training Cohort: will provide the data to be used for algorithm development and training.
  Interventions: Device: Machine-learning Algorithm
- Test or Validation Cohort: will provide data to be used for algorithm validation.
  Interventions: Device: Machine-learning Algorithm

INTERVENTIONS:
Device: Machine-learning Algorithm — System technology/Software

SUMMARY:
The study is a multi-center, prospective, non-randomized, observational study to collect data to develop and validate a machine learning algorithm for early detection of worsening heart failure events using multi-parametric sensor data from wearable data capture device The VESTA study will enroll up to 552 subjects in up to 25 centers in order to collect data on a total of at least 56 worsening heart failure events (independently adjudicated hospitalizations or unscheduled intravenous administration of decongestive drugs).The duration of follow-up per participant will be between 3-6 months.

DETAILED DESCRIPTION:
The study is an international, multicenter, prospective, open-label, non-randomized single group study, with no control group.

The study has 2 phases: the first phase is to train and develop the automated learning algorithm; the second phase is to validate the algorithm.

The participants will be assigned into two cohorts:

1. Cohort 1 will provide the data to be used for algorithm development and training.
2. Cohort 2 will provide data to be used for algorithm validation.

It has been estimated that approximately 276 subjects are required for each cohort in order to accumulate the minimum number of cases for the study's primary objective. Sequential enrolment will be implemented by regional blocks according to an estimation of the regional distribution of subjects.The sample size and regional distribution of subjects are estimates and the study is endpoint driven to achieve at least 28 WHF events with corresponding analyzable device data. Fewer subjects may be enrolled should the required number of events be acquired at a faster rate than calculated and the regional proportions of subjects may vary according to regional enrollment rates.

All participants will undergo the same study procedures, irrespective of their cohort assignment. Each subject will receive the study device kit (garment and smart phone with charger) at enrollment and will be followed up for up to 6 months, or until at least 28 worsening heart failure (WHF) events per cohort have been acquired. Even if the required number of events have been acquired, all participants will be followed up for a minimum of at least 3 months.

The study will collect data; however no data collected by the device will be made available to clinical care personnel during the study and as such no medical action will be taken based on the device. Medical follow-up will be according to standard practice as per each investigational site, which will be documented AND there will be no additional medical intervention on the study participants. The participants are required to agree to be compliant with the use of the device.

There is no masking of device allocation or procedures. However, the clinical investigators, treating physicians and the independent clinical events adjudication committee (IEAC) members will be blinded to all sensor data throughout the study.

The investigators developing the algorithm will have no access to the validation cohort database before the parameters of the algorithm have been fixed by the training cohort.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and above
* New York Heart Association(NYHA) functional class II-IV
* Reduced ejection fraction (HFrEF) with left ventricular ejection fraction (LVEF) ≤40%
* History of chronic HF as evidenced by

  * LVEF ≤40% measured at least 30 days before enrollment
  * N-terminal-pro hormone brain-type natriuretic peptide (NT-proBNP) > 500 pg/mL OR brain-type natriuretic peptide (BNP) >150 pg/mL; tested no longer than one month prior to inclusion.
* At increased risk for HF decompensation as defined by

  * currently inpatient with hospital admission due to HF decompensation (acute on chronic heart failure), or
  * history of hospitalization for HF decompensation in the last 6 months
* Understands the study requirements and the study procedures and provides written informed consent before any trial-specific tests or procedures are performed

Exclusion Criteria:

* Known allergy to any component of the study device (cotton, elastane, polyester)
* Current HF hospitalization due to acute de novo heart failure
* Current HF decompensation due to triggers like surgery or perioperative complications, pulmonary embolic episode or acute myocardial infarction
* Severe chronic kidney disease with glomerular filtration rate (GFR) <30 ml/ min/1.73 m2 and/or renal replacement therapy
* Evidence of hepatic disease as determined by any one of the following: serum glutamic-oxaloacetic transaminase (SGOT/AST) or serum glutamic-pyruvic transaminase (SGPT/ALT) values exceeding 3x upper limit of normal, bilirubin >1.5 mg/dl
* Body mass index (BMI)>35 kg/m2
* Planned surgery or other procedures within 6 months after the inclusion
* Severe uncorrected valvular heart disease, or hypertrophic obstructive cardiomyopathy, active myocarditis, constrictive pericarditis, or clinically significant congenital heart disease
* Receiving mechanical circulatory support
* Candidates on heart transplant list
* Factors or conditions, that according to investigator assessment may affect compliance with protocol or cause confound data interpretation. Examples may include but are not limited to:

  * Cardiac conditions or interventions such acute coronary syndrome, major cardiovascular surgery including coronary artery bypass graft (CABG), percutaneous coronary intervention (PCI) or implantation of a cardiac resynchronization therapy (CRT) device within 3 months prior to inclusion, or having certain implanted cardiac devices that affect cardiac condition or circulation,
  * Other serious medical illness (e.g., cancer) with estimated life expectancy of less than 12 months.
  * Current problems with substance addiction
* Participating in another investigational drug or device clinical trial
* Pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be enrolling male and female patients with history of chronic heart failure.
Sampling Method: Non-Probability Sample
Enrollment: 552 (Estimated)
Dates: Start 2021-05-31 (Estimated); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Detection of worsening heart failure (WHF) event | 6 months
  Sensitivity and Specificity of detection of WHF event by a machine-learning algorithm system using multi-parametric data captured by non-invasive telemonitoring.
  WHF event definition:
  * Any hospital admission for WHF(e.g. due to new or progressive symptoms/signs of decompensated HF including significant weight gain, worsening dyspnea or fatigue, newly elevated jugular venous pressure, new cardiac S3 gallop rhythm, the development of pulmonary rales, hepatic congestion or lower extremity edema), OR
  * Any administration of intravenous HF therapy in an unscheduled setting (e.g. clinic/office/emergency department, ED).

SECONDARY OUTCOMES:
Hospitalizations for HF that did not meet WHF | 6 months
  Algorithm System Detection of HF-associated health care utilization events not eligible to be considered as primary events
  Number of days hospitalized for HF (total number of days and per hospitalization)
HF-hospitalization in number of days | 6 months
  System Detection of HF-associated health care utilization events not eligible to be considered as primary events
  Number of days hospitalized for HF (total number of days and per hospitalization)
Outpatient health encounters leading to changes or adjustments of oral HF medication | 6 months
  Algorithm System Detection of HF-associated health care utilization events not eligible to be considered as primary events
Other healthcare encounters do not meet criteria of WHF event, points a, b and c but are deemed related to HF | 6 months
  Algorithm System Detection of HF-associated health care utilization events not eligible to be considered as primary events
Number of Adverse and Serious Adverse Events known to be associated with wearable devices with sensors | Occuring during the 6 month follow-up
  General device safety will be assessed through adverse event monitoring
Acceptability and usability of study data capture device assessed by Study Ergonomics and Usability Questionnaire | 6 months
  Patient-reported data in Ergonomics and Usability Questionnaire administered at monthly intervals.
  A Likert-like scale is used for scoring, with scores of 1-5, with higher scores signifying agreement with the questions.
Frequency and duration of study data capture device assessed by Study Frequency and duration of use Questionnaire | 6 months
  Patient-reported data in Frequency and duration of use Questionnaire administered at monthly intervals.

OTHER OUTCOMES:
All-cause hospitalizations | 6 months
  Algorithm System Detection of hospitalization events not eligible to be considered as heart failure associated events.
Deaths (Heart failure attributed) | 6 months
  Algorithm System Detection of deaths (Heart failure attributed)
Deaths (all-cause) | 6 months
  Algorithm System Detection of deaths (all cause)
Time-to-event (from alert to event) | 6 months
  Time from alert to event will be assessed for the following events to evaluate the ranges of alert to clinical event time windows for WHF events and non-HF hospitalization events

IPD SHARING:
Plan to Share IPD: No